CLINICAL TRIAL: NCT03366012
Title: The Acceptability of a Rapid Assessment of Esophageal Adenocarcinoma Risk Test (REACT)
Brief Title: Rapid Assessment of Esophageal Adenocarcinoma Risk Test
Acronym: REACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Product recall
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Julian A Abrams, MD, Associate Professor of Medicine and Epidemiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AAAR5884
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma
Keywords: Cytosponge; GERD
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cytosponge Test (Other): This arm will include individuals without formal diagnosis of Barrett's esophagus.
  Interventions: Device: Cytosponge

INTERVENTIONS:
Device: Cytosponge — The Cytosponge consists of a 3cm diameter, polyester, medical grade spherical sponge on a string, compressed within a gelatin capsule. The capsule is swallowed while the patient or the research specialist holds onto the string. After 3-5 minutes the gelatin capsule dissolves allowing the spherical sponge to expand. The sponge is then retrieved by gently pulling on the string, thus collecting cells along the passageway through the entire length of the esophagus. The sample is then put into a preservative to be processed for immunohistochemical testing for trefoil factor 3 (TFF3) to determine diagnosis of Barrett's esophagus.

SUMMARY:
This study aims to evaluate the acceptability of a new non-invasive screening device to test for Barrett's esophagus. The investigators will prospectively enroll 100 patients to undergo Cytosponge testing. The time of involvement for an individual will range from 2 weeks to 2 months, depending on the results of the Cytosponge test and time to follow up endoscopy, if indicated.

DETAILED DESCRIPTION:
The incidence of esophageal adenocarcinoma (EAC) has risen over the past half century and continues to have a dismal prognosis. Even though it has been established that Barrett's esophagus (BE) is the precursor lesion to EAC, more than 90% of EAC patients are never diagnosed with BE beforehand. Thus, the opportunity is missed to identify most patients at high risk for EAC who could benefit from surveillance and early endoscopic therapy, which in turn may lower EAC mortality. Upper endoscopy is the only means to diagnose BE, yet widespread endoscopic screening is impractical and expensive. There is an urgent need to develop minimally-invasive methods of BE screening that can be easily performed in the primary care setting to allow for efficient and cost-effective interventions to decrease EAC mortality.

ELIGIBILITY:
Inclusion Criteria:

Males:

Ages 50-75 and at least one of the following:

* Gastro-esophageal reflux disease (GERD)* or
* Family history (first degree relative) with Barrett's esophagus or esophageal adenocarcinoma or
* Both body mass index (BMI) ≥30 or
* A history of cigarette smoking (at least 10 pack years)

Females:

Ages 50-75 and GERD* and at least one of the following:

* Family history (first degree relative) with Barrett's esophagus or esophageal adenocarcinoma or
* BMI ≥30 or
* A history of cigarette smoking (at least 10 pack years)

Exclusion Criteria:

* History of gastric or esophageal cancer
* History of esophageal surgery
* Known untreated esophageal stricture or uninvestigated dysphagia
* Previous upper endoscopy within 10 years
* Cancer within 3 years except for non-melanoma skin cancer
* Portal hypertension, with or without known varices
* Uncontrolled coagulopathy
* Uncontrolled major comorbid illness
* Inability to tolerate or contraindication to upper endoscopy
* Inability to give informed consent

GERD defined as either a history of frequent heartburn or fluid regurgitation symptoms (at least weekly for 6 months) or regular use of proton pump inhibitors or histamine-2 receptor antagonists.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Abrams, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cytosponge Test
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cytosponge Test
Number analyzed (Participants) | 51
Age, Continuous [Mean (Full Range); unit: years] | 64 [50 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Participation Rate
Description: Participation rate is defined as the percent of patients who agree to undergo Cytosponge testing among number of eligible patients offered Cytosponge testing.
Time Frame: 1 Day
Measure: Number; unit: percent of participants
Arm/Group | Cytosponge Test
Number analyzed (Participants) | 51
percent of participants | 58.6

2. Primary Outcome: Patient Tolerability Determined by Score on Likert Scale
Description: After undergoing the Cytosponge test, subjects will be asked to take a "Cytosponge Post-Procedure Questionnaire" to assess tolerability using a Likert scale from 1 (no discomfort) to 10 (severe discomfort) and whether they would be willing to undergo Cytosponge testing again (yes/no). The scale for each question is rated 1 to 10. Lower scores are "better" (greater tolerability for that particular measure), higher scores are "worse" (less tolerable for that particular measure). Each question on the questionnaire will be assessed independently (i.e. one score per question). No total scores are calculated.
Time Frame: 1 Day
Population: Data was not collected due to study termination.
Arm/Group | Cytosponge Test
Number analyzed (Participants) | 0

3. Secondary Outcome: Positive Predictive Value (PPV)
Description: The PPV is the proportion of patients with endoscopic and histologic evidence of Barrett's esophagus on upper endoscopy from the total number of patients with TFF3-positive Cytosponge test who undergo a follow up endoscopy.
Time Frame: 1 Day
Population: Data was not collected due to study termination.
Arm/Group | Cytosponge Test
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Adverse Events (AEs)
Description: Total number of all AEs related to Cytosponge testing
Time Frame: 1 Day
Measure: Number; unit: study-related adverse events
Arm/Group | Cytosponge Test
Number analyzed (Participants) | 51
study-related adverse events | 0

5. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: Total number of all SAEs related to Cytosponge testing
Time Frame: 1 Day
Measure: Number; unit: serious study-related adverse events
Arm/Group | Cytosponge Test
Number analyzed (Participants) | 51
serious study-related adverse events | 0

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Cytosponge Test
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 2/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytosponge Test (N=51)
Fever (General disorders) | 1
Sore throat (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03366012/Prot_SAP_000.pdf